CLINICAL TRIAL: NCT03882190
Title: The Clinical Significance of Ovarian Function Detection and Protection in Fertility Preservation Surgery for Ovarian Malignancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAHoWMU-CR2019-07-101
Record Dates: First submitted 2019-03-17; First posted 2019-03-20 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Fertility Preservation Surgery; Ovarian Malignancy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (No Intervention)
- group 2 (Experimental)
  Interventions: Drug: GnRHa

INTERVENTIONS:
Drug: GnRHa — patients in the experimental group are supposed to receive GnRHa preoperatively and postoperatively according to their individual situation
  Arms: group 2

SUMMARY:
The design of this prospective interventional study is to investigate the clinical significance of applying GnRHa preoperatively and postoperatively and detecting physical and endocrinic change in fertility preservation surgery

DETAILED DESCRIPTION:
20 patients with ovarian maligancies are anticipated to be enrolled in this study within 2 years. With their permission, they will be randomized into the control group and the experimental group when the latter is supposed to receive GNRHa preoperatively and postoperatively. And their physical and endocrinic indexes will be monitored. The effect of extra use of GnRHa will be observed by comparing these two groups' outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in the study with informed consent;
2. Females aged 10-90 who are confirmed with ovarian malignancy and are willing to receive GnRHa experimentally to preserve their fertility function.

Exclusion Criteria:

1. Pregnancy, lactation and postmenopause;
2. Suspected or identified as other tumors of genital tract;
3. History of hyperparathyroidism, infectious diseases (tuberculosis, AIDS), autoimmune diseases, or digestive system diseases (malabsorption, crohn disease and dysentery);
4. Other diseases or heavy injuries that will interfere with the results;
5. Simultaneous participation in another clinical study with investigational medicinal product(s) or researcher thinks the subjects are not suitable for this trial.

Ages: 1 Year to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2021-03-15 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
the content of FSH(mIU/mL), LH(mIU/mL), E2(pmol/L), P(nmol/L), T(nmol/L) and PRL(nmol/L) | 1 year during the perioperative period
  by monitoring six above-mentioned hormones preoperatively and postoperatively, the ovarian function is evaluated
the volume of ovary(cm*cm*cm) | 1 year during the perioperative period
  by monitoring the change of ovarian form and volume, we evaluate the physical ovarian transformation
the ovulating period | 1 year during the perioperative period
  by comparing the ovulating period perioperatively and postoperatively between two groups, we assess the GnRHa effect on the reproductive function

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT03882190/Prot_SAP_000.pdf